CLINICAL TRIAL: NCT03374995
Title: Pilot Study: KeraStat Cream for Radiation Dermatitis
Brief Title: Topical Keratin in Treating Radiation Dermatitis in Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00046759; NCI-2017-02011 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 97417 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2017-11-29; First posted 2017-12-15 (Actual); Results first posted 2020-02-12 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2020-02

CONDITIONS: Breast Carcinoma; Radiation-Induced Dermatitis
MeSH Terms: conditions — Breast Neoplasms; Radiodermatitis | interventions — Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group I (topical keratin) (Experimental): Patients receive topical keratin topically at least BID until the end of radiation therapy (approximately 3-6 weeks).
  Interventions: Other: Quality-of-Life Assessment; Device: Topical Keratin
- Group II (standard of care) (Active Comparator): Patients receive standard of care as directed by radiation oncologist until the end of radiation therapy (approximately 3-6 weeks).
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
  Arms: Group II (standard of care)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Device: Topical Keratin — Given topically
  Other Names: KeraStat
  Arms: Group I (topical keratin)

SUMMARY:
This randomized pilot clinical trial studies how well topical keratin works in treating radiation dermatitis in patients with breast cancer. Radiation dermatitis is a skin condition that is a common side effect of radiation therapy. The affected skin becomes painful, red, itchy, and blistered. Topical keratin may help to improve skin appearance and hydration in patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine a preliminary estimate of the improvement of skin's natural barrier, decrease of dehydration, and reduction in the appearance of inflammation associated with radiation therapy (RT) skin toxicity as well as patients' satisfaction with their skin after the application of the medical device topical keratin (KeraStat Cream) during RT in breast cancer patients.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive topical keratin topically at least twice daily (BID) until the end of radiation therapy (approximately 3-6 weeks).

GROUP II: Patients receive standard of care as directed by radiation oncologist until the end of radiation therapy (approximately 3-6 weeks).

After completion of study treatment, patients are followed up at 4-6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast cancer, received chemotherapy, and scheduled to receive 4 to 6 weeks of radiation therapy (radiation protocol of 42 Gy+)
* Area to be irradiated representing 1-10% of total body surface area (TBSA)
* Able and willing to sign protocol consent form
* Able and willing to document symptoms and treatment details as often as needed, not to exceed daily notes
* Able and willing to have photographs of the affected area taken regularly

Exclusion Criteria:

* Women who are pregnant, lactating/nursing or plan to become pregnant
* Previous radiation therapy to the area to be treated with radiation therapy
* Receiving palliative radiation therapy
* Unhealed or infected surgical sites in the irradiation area
* Patients undergoing cytotoxic chemotherapy or concurrent Herceptin as part of overall treatment plan (tamoxifen/aromatase inhibitor allowed)
* Use of oral corticosteroids or topical corticosteroids in the irradiation area
* Use of Erbitux
* Autoimmune disease
* Skin disease in target irradiation area
* Smoker
* Known allergy to the standard of care or ingredients in KeraStat Cream

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Winkfield, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group I (Topical Keratin) | Group II (Standard of Care)
Started | 13 | 12
Completed | 13 | 11
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I (Topical Keratin) | Group II (Standard of Care) | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.15 (9.5) | 65.36 (7.18) | 62.0 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 11 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 11 | 9 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Early Adverse Skin Reactions (EASRs)
Description: The Modified ONS Criteria for Radiation-Induced Acute Skin Toxicity will be used for classification of EASRs related to the skin. Participants will report in a total of 7 visits any experience with Grade I (faint or dull erythema; dry desquamation or Grade II (tender or bright erythema, patchy, moist desquamation) acute radiation dermatitis using the RTOG (Radiation Therapy Oncology Group) grading system with Grade II considered the worse outcome. Comparative effectiveness will include the number or study participants in each arm that experience RTOG Grade I or Grade II radiation dermatitis and moist desquamation.
Time Frame: Up to 4 weeks post-RT
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Topical Keratin) | Group II (Standard of Care)
Number analyzed (Participants) | 13 | 11
Participants
  Grade I Acute Radiation Dermatitis | 13 | 10
  Grade II Acute Radiation Dermatitis | 4 | 6
  Moist Desquamation | 1 | 0

2. Primary Outcome: Change in Quality of Life
Description: A 10-item assessment completed at each visit (7 total) to measure participant's Dermatology Life Quality Index. Score range is 0-3 (very much = 3; a lot = 2; a little = 1; and not at all or not relevant = 0) Maximum score of 30. The higher the score the more qualify of life is impaired. The average DQLI score at each study visit will be compared between the KeraStat® Cream arm and the SOC arm as a study effectiveness measure.
Time Frame: Baseline to up to 7 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group I (Topical Keratin) | Group II (Standard of Care)
Number analyzed (Participants) | 13 | 11
score on a scale
  Visit 1 (baseline) | 0.31 (0.82) | 2.73 (5.26)
  Visit 2 | 0.77 (1.31) | 1.64 (2.06)
  Visit 3 | 2.23 (3.85) | 1.91 (2.11)
  Visit 4 | 2.85 (2.98) | 2.36 (2.53)
  Visit 5 | 4.75 (6.99) | 5.27 (5.01)
  Visit 6 | 4.25 (4.87) | 6.18 (5.70)
  Visit 7 | 0.85 (1.10) | 1.00 (2.05)

3. Primary Outcome: Physician Observed Improvement in Skin Appearance
Description: Skin appearance was assessed by the treating physician at each visit (total of 7) using the Radiation Therapy Oncology Group (RTOG) Toxicity scale Grade 1 and Grade 2 assessed only. Score = (Grade 1 (follicular, faint or dull erythema, dry desquamation and Grade 2 (tender or bright erythema, patchy, ,moist desquamation) with Grade 2 being the worst for this study. Scores range from 0 to 2, with higher values being the worst. The average RTOG score at each study visit will be compared between the KeraStat® Cream arm and the SOC arm as a study effectiveness measure.
Time Frame: Baseline to up to 7 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group I (Topical Keratin) | Group II (Standard of Care)
Number analyzed (Participants) | 13 | 11
units on a scale
  Visit 1 (baseline) | 0.00 (0) | 0.00 (0)
  Visit 2 | 0.15 (0.36) | 0.09 (0.29)
  Visit 3 | 0.62 (0.49) | 0.55 (0.50)
  Visit 4 | 1.00 (0.68) | 0.82 (0.38)
  Visit 5 | 1.17 (0.55) | 1.00 (0.43)
  Visit 6 | 1.00 (0) | 1.36 (0.64)
  Visit 7 | 0.23 (0.42) | 0.30 (0.46)

4. Primary Outcome: Number of Participants Reported Change in Skin Appearance Using the Dermatology Quality of Life Index Scale
Description: Change in skin appearance by the participants' self-report using the Dermatology Quality of Life Index (DLQI) was used to assess skin after completion of radiation. Score range is 0-3 (very much = 3; a lot = 2; a little = 1; and not at all or not relevant = 0) Maximum score of 30. A higher score shows better performance/improvement in skin appearance. The average Dermatology Qualify of Life Index score each study visit will be compared between the two arms with the number of participants reporting a score.
Time Frame: Baseline to up to 7 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Group I (Topical Keratin) | Group II (Standard of Care)
Number analyzed (Participants) | 13 | 11
Participants
  Visit 1 (baseline) | 2 | 4
  Visit 2 | 6 | 6
  Visit 3 | 8 | 8
  Visit 4 | 11 | 7
  Visit 5 | 11 | 10
  Visit 6 | 10 | 10
  Visit 7 | 7 | 2

ADVERSE EVENTS:
Time Frame: Up to 30 days post radiation therapy
Description: Expected side effects of radiation therapy that occurred at expected timeframes and severity (e.g., erythema, edema, desquamation) were not considered to be adverse events.
Arm/Group | Group I (Topical Keratin) | Group II (Standard of Care)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 0/13 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT03374995/Prot_SAP_000.pdf